CLINICAL TRIAL: NCT06519682
Title: U-R-Immune Glioma (CA209-1245): A Pilot Study Investigating Upfront Adaptive Immunotherapy Approach in Children, Adolescent and Young Adult (CAYA) Patients With Replication-Repair Deficient (RRD) High-Grade Gliomas (HGG)
Brief Title: A Pilot Study Investigating Upfront Adaptive Immunotherapy Approach in Children, Adolescent and Young Adult (CAYA) Patients With Replication-Repair Deficient (RRD) High-Grade Gliomas (HGG)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Daniel Morgenstern (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Anti Cancer Fund (Unknown)
Responsible Party: Sponsor-Investigator, Daniel Morgenstern, Senior Medical Officer, The Hospital for Sick Children
Organization: The Hospital for Sick Children (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U-R-Immune Glioma (CA209-1245)
Record Dates: First submitted 2024-07-16; First posted 2024-07-25 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: High Grade Glioma; Replication Repair Deficient
MeSH Terms: conditions — Glioma | interventions — Nivolumab; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Domain 1 - Upfront ICI (Active Comparator): Initially 12 eligible patients will be enrolled for upfront ICI. At 12 week assessment if >6 patients have response (NO radiation for recurrence/progression), an additional 6 patients will be enrolled for upfront ICI. All patients will be assessed at 12 weeks from the start of ICI. If 6 or fewer patients have response (NO radiation for progression/recurrence), no more patients will be recruited to this domain.
  Interventions: Drug: Nivolumab
- Domain 2 - Radiation + ICI → maintenance ICI (Active Comparator): All the patients experiencing tumor progression on domain 1 will be eligible for domain 2 and will receive a combination of radiation and nivolumab followed by maintenance nivolumab for 2 years. To be eligible for domain 2 post recurrence patients will need surgery/biopsy at recurrence. If 6 RRD-glioblastoma will recur/progress at 12 weeks on domain 1 then 8 additional eligible patients may be directly enrolled in domain 2.
  Interventions: Drug: Nivolumab; Radiation: Radiation

INTERVENTIONS:
Drug: Nivolumab — All patients will be administered Nivolumab with or without radiation
Radiation: Radiation — Radiation
  Arms: Domain 2 - Radiation + ICI → maintenance ICI

SUMMARY:
This is open label, multicentre, single arm, pilot study of upfront nivolumab in patients with RRD-glioblastoma with favorable immune/genomic biomarkers. The purpose of the study is to use upfront immune checkpoint inhibitor (ICI) to delay/avoid radiation for patients with RRD-glioblastoma with favorable clinical (Gross total resection (GTR) or near total resection (NTR)) and biological (RRD, hypermutation, immune activation) biomarkers. At progression, patients will be undergoing surgery/biopsy and will get a combination of radiation + ICI followed by maintenance ICI. This model will allow us to additionally study the evolution tumor in response to ICI. The study will have two domains.

DETAILED DESCRIPTION:
Domain 1 - Upfront ICI Initially 12 eligible patients will be enrolled for upfront ICI. At 12 weeks assessment if >6 patients have response (NO radiation for progression/recurrence), an additional 6 patients will be enrolled for upfront ICI. Nivolumab will be administered at a dose of 6 mg/kg every 4 weeks (cycle). All patients will be assessed at 12 weeks (3 cycles) from the start of ICI. If 6 or more out of 12 RRD-glioblastoma will recur/progress, no more patients will be recruited to this domain.

Domain 2 - Radiation + ICI → maintenance ICI All the patients experiencing tumor progression on domain 1 will be eligible for domain 2 and will receive a combination of radiation and nivolumab followed by maintenance nivolumab for a total of 2 years (24 cycles). To be eligible for domain 2 post recurrence patients will need surgery/biopsy at recurrence. If 6 RRD-glioblastoma will recur/progress at 12 weeks on domain 1 then 8 additional eligible patients may be enrolled directly in domain 2.

Patients may receive up to a total of approximately 2 years of treatment (up to 24 cycles). Follow-up may continue for up to one year following treatment discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* 3.1.1 Age: Patients must be ≥12 months and ≤25 years of age at the time of signing informed consent/assent.

3.1.2 Diagnosis: Patients must have a histologically confirmed diagnosis of glioblastoma.

3.1.3 Proof of RRD: By tumor immunohistochemistry showing functional loss of mismatch repair gene expression (MLH1, MSH2, MSH6, PMS2), or based on prior germline testing confirming congenital mismatch repair deficiency (CMMRD) or Lynch syndrome. To be done locally. Results have to be available within four weeks of last surgery.

3.1.4 Tumor Tissue Specimen: Provide a tumor tissue specimen for molecular profiling, including TMB analysis. Any tumor sequencing data if available at time of enrolment will be recorded for relevant pathogenic variants in the mismatch repair and polymerase-proofreading genes to suggest RRD. A specimen from the time of relapse/ progression while on the study is required as well, when applicable.

3.1.5 Favorable immune markers: High PD1 and CD8 positivity as detailed in the lab manual. To be done locally. Results have to be available within 4 weeks of last surgery.

3.1.6 Surgical and disease status: Patients should have had Gross total resection (GTR)/Near Total Resection (NTR) as confirmed by the post-surgery scan. Patients are allowed a second look surgery to achieve NTR/GTR provided no tumor directed systemic or radiation therapy has been administered before this second surgery. Patients should be able to start therapy within 4 weeks of last surgery.

3.1.7 Allowable Prior Therapy: 3.1.7.1 Patients must have recovered from the acute toxic effects of all prior anti-cancer therapies (with the exception of alopecia and lymphopenia). Previous treatment with nivolumab and/or other anti- PD-1/PD-L1 inhibitors for other prior tumors (other than high-grade glioma) will be permitted.

3.1.7.2

Prior Therapy: No prior therapy except surgery will be permitted for high grade glioma. If the patient was previously diagnosed and treated for another tumor (other than high grade glioma), the patients must have completed that treatment and have no active disease in order to be enrolled in this trial The following time periods apply for prior therapy for other tumors:

* Cytotoxic chemotherapy: At least 21 days prior to initiation of protocol therapy from the last dose of cytotoxic or myelosuppressive chemotherapy; at least 42 days if prior nitrosourea (such as lomustine, CCNU).
* Hematopoietic growth factors: At least 7 days prior to initiation of protocol therapy from the last dose of short-acting growth factor; at least 14 days for long-acting.
* Anti-cancer agents not known to be myelosuppressive: At least 7 days prior to initiation of protocol therapy from the last dose.
* Interleukins, interferons, and cytokines (other than hematopoietic growth factors): At least 21 days prior to initiation of protocol therapy from the last dose.
* Antibodies: At least 21 days prior to initiation of protocol therapy from the last dose and toxicity related to prior antibody therapy must be recovered to Grade ≤1.
* Radiotherapy: At least 14 days prior to initiation of protocol therapy from local radiotherapy; at least 150 days from total body irradiation (TBI), craniospinal radiotherapy, or radiation to

  ≥50% of the pelvis; at least 42 days from other substantial bone marrow radiation.
* Radiopharmaceutical therapy (e.g., 131I-MIBG): At least 42 days prior to initiation of protocol therapy from systemically administered radiopharmaceutical therapy.
* Autologous stem cell infusion including boost infusion: At least 42 days prior to initiation of protocol therapy.
* Cellular therapy: At least 42 days prior to initiation of protocol therapy from any type of cellular therapy.

3.1.8 Performance Status: Lansky play score ≥50 if ≤16 years of age; Karnofsky performance scale ≥50 if >16 years of age. See Appendix A. Patients unable to walk due to paralysis but who are using a wheelchair will be considered ambulatory for the purpose of assessing the performance score.

3.1.9 Organ Function: 3.1.9.1

Adequate bone marrow function defined as:

* peripheral absolute neutrophil count (ANC) ≥750/mm3 (0.75x109/L)
* platelet count ≥75,000/mm3 (75x109/L), transfusion independent, defined as not receiving platelet transfusions at least 7 days prior to initiation of protocol therapy 3.1.9.2

Adequate renal function defined as:

-creatinine clearance or radioisotope GFR ≥60 mL/min/1.73 m2; OR serum creatinine based on age/gender 3.1.9.3

Adequate liver function defined as:

* bilirubin (sum of conjugated and unconjugated) ≤1.5 x upper limit of normal (ULN) for age
* ALT (SGPT) ≤135 U/L (i.e., 3 x ULN). For the purposes of this study, the ULN for ALT (SGPT) is 45 U/L 3.1.9.4

Adequate pulmonary function defined as:

-no evidence of dyspnea at rest, no exercise intolerance due to pulmonary insufficiency, and pulse oximetry ≥92% while breathing room air 3.1.9.5

Adequate cardiac function defined as:

* no signs or symptoms of heart failure in a patient who has no history of congestive heart failure, no prior exposure to cardiotoxic drugs, and no radiotherapy to the heart; OR
* shortening fraction of ≥27% or ejection fraction of ≥50% by echocardiogram 3.1.9.6

Adequate pancreatic function defined as:

-serum lipase ≤ ULN at screening 3.1.9.7

Viral Infection:

* Human immunodeficiency virus (HIV): Infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months prior to initiation of protocol therapy are eligible.
* Hepatitis B virus (HBV): Patients with evidence of chronic infection with undetectable viral load are eligible. Suppressive therapy, if indicated, is allowed.
* Hepatitis C virus (HCV): Infected patients currently on treatment with undetectable viral load are eligible. Patients with a history of infection must have been treated and cured.

Note: Routine screening for HBV, HCV or HIV status prior to enrollment is not required.

3.1.9.8 Informed Consent: All patients and/or their parents or legally authorized representatives must have the ability to understand and the willingness to sign, provide a thumbprint (e.g.., for illiterate patients), or use an authorized method to duly document the informed consent in line with the local IRB/IEC requirements and the regulations in force). Assent, where appropriate, will be obtained according to local regulations.

Exclusion Criteria:

* 3.2.1

Concomitant Medications:

* Corticosteroids: Patients requiring systemic corticosteroids or other forms of immunosuppressive therapy within 7 days prior to initiation of protocol therapy are not eligible.
* Following initiation of protocol therapy, systemic corticosteroids or other forms of immunosuppressive therapy are permitted if administered for the treatment of toxicity, tumor flare, or pseudo-progression and can be tapered. In most cases protocol therapy must be held until the dose is tapered to 10 mg/day prednisone or equivalent. The Protocol Principal Investigator must be consulted prior to resuming treatment.
* Physiologic corticosteroids up to 5 mg/day prednisone or equivalent are permitted.
* Topical, ocular, intra-articular, intra-nasal, and inhaled corticosteroids are permitted.
* Patients with CNS tumors receiving steroids must be able to discontinue these at least 7 days prior to initiation of protocol therapy.
* Anti-cancer agents: Patients who are currently receiving other anti-cancer agents are not eligible.
* Other investigational agents: Patients who are currently receiving or have received any other investigational agent within 14 days prior to initiation of protocol therapy are not eligible.

3.2.2

CNS Tumor Bulk: Patients with CNS tumors with any of the following characteristics on imaging are not eligible:

* Tumor with any evidence of uncal herniation or mass effect leading to severe midline shift
* Tumor that in the opinion of the local investigator, shows significant mass effect after initial surgery or after second-look surgery.

3.2.3 Uncontrolled Intercurrent Illness: Patients with uncontrolled intercurrent illness including, but not limited to, ongoing active infection, symptomatic congestive heart failure (New York Heart Association Class III or IV), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements are not eligible.

3.2.4 Pregnant and/or Breastfeeding: The study agents have the potential for teratogenic or abortifacient effects. Females of reproductive potential must have a negative serum pregnancy test within 72 hours prior to initiation of protocol therapy. Additional pregnancy tests (serum or urine) should be obtained during study participation in accordance with local standards and guidelines.

Males or females of reproductive potential may not participate unless they have agreed to use an effective method of contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of treatment, and as follows:

●Females receiving nivolumab must continue an effective method of contraception for a period of 5 months after the last dose of nivolumab.

Should a female patient become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform the investigator immediately.

Due to the unknown but potential risk for AEs in nursing infants secondary to treatment of the mother with the study agents, breastfeeding must be discontinued if the mother is treated on study.

Note: Females of reproductive potential are defined as those who are past the onset of menarche and are not surgically sterile (i.e., bilateral salpingectomy, bilateral oophorectomy, or complete hysterectomy).

3.2.5 Autoimmune Disease: Patients with a history of autoimmune disease (such as autoimmune thyroid disease or inflammatory bowel disease) that has required systemic treatment within 2 years prior to initiation of protocol therapy are not eligible.

* Asymptomatic laboratory abnormalities (e.g., ANA, rheumatoid factor, altered thyroid studies) will not render a patient ineligible in the absence of a diagnosis of an autoimmune disorder.
* Patients with atopy-related conditions such as asthma, allergic rhinitis, or atopic dermatitis are not excluded.
* Replacement therapy (e.g., thyroxine, insulin, or physiological corticosteroid replacement therapy) is not considered a form of systemic treatment.

3.2.6 Interstitial Lung Disease: Patients with history of interstitial lung disease or pneumonitis are not eligible.

3.2.7 Transplant: Patients who have received previous solid organ transplant or allogenic stem cell transplant are not eligible.

3.2.8 Adverse Reaction to Study Agent(s): Patients with previous Grade 4 life-threatening reaction or other adverse reaction that in the opinion of the investigator would preclude retreatment with nivolumab, and/or other PD-1/PD-L1 antibodies are not eligible.

3.2.9 Compliance: Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible.

3.2.10 Treatment Start: Patients unable to start study protocol treatment within 14 days from the enrollment date or within 4 weeks of surgery (whichever is earlier).

3.3 Specific Criteria for Domain 2 3.3.1 Proceeding from Domain 1 to Domain 2 For patients already enrolled on the study, the following exclusion criteria specifically apply prior to proceeding to Domain 2.

3.3.1.1 Specific Exclusion Criteria

* Surgery: Patient who cannot have surgery/biopsy at recurrence/progression on Domain 1 will be discontinued from the study.
* CNS Tumor Bulk: Patients with CNS tumors with any of the following characteristics on imaging post-surgery/biopsy at progression/recurrence on Domain 1 are not eligible:

  * Tumor >= 5cm in the longest dimesion.
  * Tumor with any evidence of uncal herniation or mass effect leading to severe midline shift
  * Tumor that in the opinion of the local investigator, shows significant mass effect

Ages: 12 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
To evaluate Radiation-free survival (RFS) from start of immunotherapy | 2 years
  Radiation-free survival defined as time from start of immunotherapy to date of onset of radiation for progression/recurrence as determined by the iRANO criteria.

SECONDARY OUTCOMES:
To evaluate overall survival (OS) | 5 years
  Defined as the time from date of enrollment until death from any cause.
To evaluate progression free survival (post first progression) | 2 years
  Defined as time from first progression (post upfront ICI) to second progression as determined by the iRANO criteria.
To evaluate clinical benefit rate (CBR) | 2 years
  The proportion of patients who have no evidence of progression for at least two protocol reassessment periods as determined by the iRANO criteria.
Quality of life as measured by a validated PedsQL, generic module and PROMIS. | 2 years
  Patients and/or caregivers will complete questionnaires during regular clinic visits at three required time points: time of study enrollment, 12 weeks of therapy, end of study.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Morgenstern, MD, Study Director — The Hospital for Sick Children
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No